CLINICAL TRIAL: NCT05668273
Title: The Effect of Simulation in the Teaching of Auscultation Skills on Patient Assessment, and Anxiety and Self-Confidence With Clinical Decision Making
Brief Title: Patient Assessment, and Anxiety and Self-Confidence With Clinical Decision Making in Auscultation Skills With Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GaziU-SBF-SA-2
Record Dates: First submitted 2022-12-12; First posted 2022-12-29 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Self-Confidence
Keywords: Simulation; Nursing; Auscultation; Patient assessment
MeSH Terms: conditions — Anxiety Disorders | interventions — Educational Status; Control Groups

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental design.
Masking Description: The analysis of the tests data will be done by the statistician. No information will be given to the statistician about which group the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- education with simulated patient (Experimental): Participants will be given training on auscultation skills with a simulated patient.
  Interventions: Other: education with simulated patient
- education with simulator (Experimental): Participants will be given training on auscultation skills with a simulation.
  Interventions: Other: education with simulator
- control group (Active Comparator): Participants will be given training on auscultation skills with their peer students.
  Interventions: Other: control group

INTERVENTIONS:
Other: education with simulated patient — Students in the education with the simulated patient group will practice auscultation skills on the simulated patient with heart, lung, and bowel sounds. There will be a lecturer at the head of the group who will provide the necessary coordination. A debriefing session will be held with the students by the educator right after the students have finished the application.
  Arms: education with simulated patient
Other: education with simulator — Students in the simulator group will practice auscultation skills on high fidelity simulator with heart, lung, and bowel sounds. There will be a lecturer at the head of the group who will provide the necessary coordination. A debriefing session will be held with the students by the educator right after the students have finished the application.
  Arms: education with simulator
Other: control group — Students in the control group will practice auscultation skills on their peers with heart, lung, and bowel sounds. There will be a lecturer at the head of the group who will provide the necessary coordination.
  Arms: control group

SUMMARY:
This research is a randomized controlled experimental design. This research will be applied within the scope of the Health Assessment Course. The population of the research will be the students enrolled in the Health Assessment Course (n=138). The sample will consist of students who volunteered to participate in the research.

Introductory Specifications Form, Nursing Anxiety and Self-Confidence with Clinical Decision-Making scale, Auscultation of Heart, Lung, and Bowel Sounds Checklist, and Opinions of Students about the Auscultation Skills Training will be used in the implementation of the research.

Permission was obtained from the Gazi University Ethics Committee and the Dean of the Faculty of Health Sciences to conduct the research. Informed consent will be obtained from the students who will participate in the research.

DETAILED DESCRIPTION:
This research will be applied within the scope of the Health Assessment Course in Gazi University Faculty of Nursing in the fall and spring semesters of the 2022-2023 academic year. The population of the research will be the students enrolled in the Health Assessment Course (n=138). The sample will consist of students who volunteered to participate in the research.

Introductory Specifications Form, Nursing Anxiety and Self-Confidence with Clinical Decision-Making scale, Auscultation of Heart, Lung, and Bowel Sounds Checklist, and Opinions of Students about the Auscultation Skills Training will be used in the implementation of the research.

The researcher will teach all students the theoretical content of the subject. The students who meet the criteria for inclusion in the research will then be given the Introductory Specifications Form and the Nursing Anxiety and Self-Confidence with Clinical Decision-Making scale (pre-test). Students will be divided into three groups based on their academic averages and scale scores using stratified randomization. Students in experimental group 1 will be trained with a standardized patient, students in experimental group 2 will be trained with a high-fidelity simulator, and students in the control group will be trained with their peers. Following the completion of the application, the students will participate in a debriefing session. Students will be evaluated using checklists one week after submitting their applications. At this point, students in experimental group 1 will practice auscultation of heart, lung, and bowel sounds on a standardized patient, students in experimental group 2 will practice on a high-fidelity simulator, and students in the control group will practice on their peers.

While the students are applying, the observers will fill out the checklist for each item from the "observed," "incorrect/incomplete," and "not observed" options. Following the application, students will complete the Nursing Anxiety and Self-Confidence with Clinical Decision-Making scale (post-test).

During the spring semester, students will participate in clinical practice at various clinics two days per week as part of the Surgical Nursing Course. They also use auscultation skills in clinical settings. Students in the Experimental 1, Experimental 2, and Control groups will complete the Nursing Anxiety and Self-Confidence with Clinical Decision-Making scale and Opinions of Students about the Auscultation Skills Training at the end of the spring semester (when clinical applications are completed) (follow-up test).

Permission was obtained from the Gazi University Ethics Committee and the Dean of the Faculty of Health Sciences to conduct the research. Informed consent will be obtained from the students who will participate in the research.

The quantitative data from this study will be digitized in the SPSS package program, and the necessary statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Enrolling in the Health Assessment Course for the first time
* Volunteering to participate in research

Exclusion Criteria:

* Having a high school, associate, or undergraduate degree in a health-related field,
* Take a previous course in health assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
The Change of the Nursing Anxiety and Self-Confidence with Clinical Decision-Making | 5 months
  This scale consists of 27 questions. Separate scores are obtained for self-confidence and anxiety from the scale. For both self-confidence and anxiety sections of the scale; It has three sub-dimensions: "Using resources to obtain information and listening fully (13 questions)", "Using the information at hand to determine the problem (7 questions)" and "knowing and acting (7 questions)". As the scores obtained from the self-confidence section and its sub-dimensions increase, the self-confidence level of the student increases, and the low scores obtained from the anxiety section and its sub-dimensions indicate a low level of anxiety. In the scale prepared in a six-point likert type; The lowest score that can be obtained from the self-confidence and anxiety sections is 27, and the highest score is 162.
Auscultation of Heart, Lung and Bowel Sounds Checklist | One week
  The checklist has been prepared in line with the objectives of the course content on heart, lung and bowel sounds. It consists of application steps that include the process steps in detail. It was created in the form of a rubric in order to observe the students objectively. Each item in the checklist has different scores according to its importance. The total score to be taken from all of them is 50. Expert opinion of the checklist was taken by 5 faculty members who are experts in the field.

SECONDARY OUTCOMES:
Opinions of students about the auscultation skills training | one week
  The form will be used in order to learn the reflection of auscultation skills education in clinical practice. The interview questions in the form were created in line with the academic experiences of the researchers. The interview form consists of 3 open-ended questions: 1) how the training affected their feelings and thoughts in clinical practice, 2) how it affected their application of physical examination skills for the patients they care for in the clinic, and 3) what would have changed if you had gone to the clinic without this training. This form will be evaluated by thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Nurcan Çalışkan, Prof., Study Director — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Bektaş, İ., Yardımcı, F., Bektaş, M., & White, K. A. (2017). Psychometric properties of the Turkish version of nursing anxiety and self-confidence with clinical decision-making scale (NASC-CDM-T). Dokuz Eylül Üniversitesi Hemşirelik Fakültesi Elektronik Dergisi, 10(2), 83-92.
- [Background] Gawlik, K.S., Melnyk, B.M., Teall, A.M. (Eds.), (2022), Evidence-based physical examination handbook, Springer Publishing Company, LLC
- [Background] Hogan-Quigley, B., Palm, M.L., Bickley, L.S., (2012). Bates' nursing guide to physical examination and history taking. Wolters Kluwer Health | Lippincott Williams & Wilkins.